CLINICAL TRIAL: NCT05901558
Title: Strategies for Toddler ASD With Remote-therapy (STAR) Model for Early ASD Toddlers: a Randomized Trial
Brief Title: Strategies for Toddler ASD With Remote-therapy (STAR) Model for ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAR-ASD 1.0
Record Dates: First submitted 2023-05-11; First posted 2023-06-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Therapy
Keywords: Autism; Naturalistic developmental behavioral intervetion; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAR intervention group (Experimental): The intervention strategies in STAR model are designed under the Naturalistic Developmental Behavioral Intervention (NDBI) framework which are implemented in natural settings targeting at improving social and communicational capabilities. The structure of the STAR model is with 2 modules and 16 sessions. Module I derives from our previous offline parent-tutoring courses with 8 intervention strategy topics combining academic instruction and real child demonstration but modified into on-line version. Module II is designed specifically for long-term consolidation of parents' intervention skills containing 8 biweekly sessions of distance coaching with parents practicing intervention with their children in real time at home.
  Interventions: Behavioral: Strategies for Toddler ASD with Remote-therapy (STAR)
- community intervention group (Other): This group will have community interventions parents can choose.
  Interventions: Behavioral: Community intervention

INTERVENTIONS:
Behavioral: Strategies for Toddler ASD with Remote-therapy (STAR) — The intervention strategies in STAR model are designed under the Naturalistic Developmental Behavioral Intervention (NDBI) framework which are implemented in natural settings targeting at improving social and communicational capabilities
  Arms: STAR intervention group
Behavioral: Community intervention — Regular community intervention
  Arms: community intervention group

SUMMARY:
The project aims to develop and implement the Strategies for Toddler Autism spectrum disorder(ASD) with Remote-therapy (STAR) model for early toddlers with ASD in local community sites in Shanghai. It's a randomized control trial lasting 3 years. The children will be divided into 2 groups, one for STAR intervention group and the other for community intervention group. The STAR intervention group will be performed STAR other than community intervention.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) brings enormous economic and emotional burdens to families and society with its ever-increasing prevalence. Early intervention has been proved as the key treatment to ASD. Along with increasing number of ASD children identified and diagnosed at early stage, the needs for effective early intervention are dramatically increasing. Though therapist-delivered intensive programs for toddlers yield substantive developmental gains, they tend to be costly and with extremely limited resource. The lockdowns during the COVID-19 pandemic brings even more obstacles for the children and families to get access to the resource of intervention. As such, the traditional intervention models are not fit for wide implementation within the Chinese public health systems and pandemic situation.

To solve this dilemma, this project aims to develop and implement the Strategies for Toddler ASD with Remote-therapy (STAR) model for early toddlers with ASD in local community sites in Shanghai. To maximize the intervention effect, the intervention strategies in STAR model are designed under the Naturalistic Developmental Behavioral Intervention (NDBI) framework which are implemented in natural settings targeting at improving social and communicational capabilities. The structure of the STAR model is with 2 modules and 16 sessions. Module I derives from our previous offline parent-tutoring courses with 8 intervention strategy topics combining academic instruction and real child demonstration but modified into on-line version. Module II is designed specifically for long-term consolidation of parents' intervention skills containing 8 biweekly sessions of distance coaching with parents practicing intervention with their children in real time at home.

ELIGIBILITY:
Inclusion Criteria:

* Children screened as positive for ASD.
* Two-tiered screening process combing Level 1(The Modified Checklist for Autism in Toddlers-Revised/Follow-Up , M-CHAT-R/F) and Level 2 (The Screening Tool for Autism in Toddlers and Young Children, STAT)

Exclusion Criteria:

* Other neurologic or degenerative diseases;
* Severe hearing or visual impairment;
* Genetic anomaly which may affect impact on intervention;
* Not available for regular intervention and follow-up.

Ages: 16 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Communication and Symbolic Behavior Scales Developmental Profile（CSBS） | from enrollment (T0) to 1 year(T2)
  The Checklist consists of 24 questions that range from 2 to 4 points within each of 7 Clusters, including language predictors: emotion and eye gaze, communication, gestures, sounds, words, understanding, and object use. Give credit of 0 points for items checked Not Yet, 1 point for items checked Sometimes, or 2 points for items checked Often. 7 Cluster scores will be summed to yield three Composite scores (including expressive speech, symbolic and communication) and a total score. The change of each score for T0, T1 and T2 will be measured.

SECONDARY OUTCOMES:
Autism Diagnostic Observation Schedule-Second edition(ADOS-2) | from enrollment (T0) to 1 year(T2)
  Autism Diagnostic Observation Schedule-Second edition(ADOS-2):
  The results from the social affect(SA) and restricted and repetitive behavior (RRB, subdomains were added together to generate the total raw score. The total raw score was converted into the ADOS calibrated severity score , ranging from 1 to 10, with 10 being the most severe.
Parenting Stress Index/Short Form （PSI/SF） | from enrollment (T0) 1 year(T2)
  3 sub-scales, including parent distress (PD), parent-child dysfunctional interaction(PCDI), difficult child (DC). This scale assesses stress in parents.
The Griffiths Mental Development Scales (GMDS) | from enrollment (T0) 1 year(T2)
  GMDS includes six subscales:
  Locomotor (Lm), Personal and Social (P/S), Hearing and Speech (H/Sp), Eye and Hand (E/Hd), Performance (Pf) and Practical Reasoning (Pr). The raw scores were transformed into developmental quotients (DQ) using the standard method.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No